CLINICAL TRIAL: NCT03821857
Title: Sex-Specific Effects of Endocrine Disruption on Aging and Alzheimer's Disease
Acronym: SEED-AD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kejal Kantarci, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-008476; U54AG044170-09 (NIH); R01AG093767 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Women (Experimental): 18F-Flortaucipir and 11C-Pittsburgh compound-B radioligands will be used for experimental PET imaging of beta-amyloid and neurofibrillary tau pathology
  Interventions: Drug: 18-F-Flortaucipir

INTERVENTIONS:
Drug: 18-F-Flortaucipir — Radioligands for PET imaging of beta-amyloid and neurofibrillary tangle tau pathology
  Other Names: 11C-Pittsburgh Compound-B

SUMMARY:
The researchers are trying to determine whether ovarian hormones are associated with aging processes and with the risk of developing Alzheimer's disease in women.

DETAILED DESCRIPTION:
The proposed project will enroll a total of 614 women.

Mayo Clinic Rochester Participants: Each women will have 2-3 clinic visits consisting of cognitive testing, tests of physical function, questionnaires, and a blood draw. All women will also undergo clinical neuroimaging, which includes structural MRI, β-amyloid (Aβ) deposition on PET as a biomarker of Aβ pathology, and tau deposition on PET as a marker of neurofibrillary tangles using AV-1451. All participants will have previously participated and will return by invitation only.

Mayo Clinic Jacksonville Participant: Only African American Women will be enrolled at this site. Each women will have 1-3 clinic visits consisting of physical function testing and neuroimaging, which includes structural MRI, β-amyloid (Aβ) deposition on PET as a biomarker of Aβ pathology, and tau deposition on PET as a marker of neurofibrillary tangles using AV-1451.

ELIGIBILITY:
Mayo Clinic Rochester-

Inclusion Criteria:

* Women who previously participated in this study
* Currently aged 60 years and older
* More than six months post chemotherapy or major surgery requiring general anesthesia
* Willing and able to sign informed consent

Exclusion Criteria:

* Not able to read and speak English
* In hospice
* Claustrophobic
* If undergoing Tau imaging, cannot have QT Prolongation

Mayo Clinic Jacksonville-

Inclusion Criteria:

* African American Women
* Currently aged 60 years and older
* More than six months post chemotherapy or major surgery requiring general anesthesia
* Willing and able to sign informed consent

Exclusion Criteria:

* Not able to read and speak English
* In hospice
* Claustrophobic
* If undergoing Tau imaging, cannot have QT Prolongation

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 614 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
18F-Flortaucipir PET imaging | 1 day
  Cortical 18F-Flortaucipir PET imaging measured once in each participant
Pittsburgh compound-B PET imaging | 1 day
  Global cortical SUVR measured once in each participant

CONTACTS AND LOCATIONS:
Overall Officials: Kejal Kantarci, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No